CLINICAL TRIAL: NCT03625986
Title: Does Switching to Nicotine Containing Electronic Cigarettes Reduce Health Risk Markers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Jonathan Foulds, Professor, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 8948; U01DA045517 (NIH)
Record Dates: First submitted 2018-08-02; First posted 2018-08-10 (Actual); Results first posted 2025-03-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Tobacco Dependence
Keywords: smoking; electronic cigarettes; nicotine; ecig
MeSH Terms: conditions — Tobacco Use Disorder; Smoking; Vaping

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nicotine-Containing Electronic Cigarette (Experimental): The experimental group will be provided with and encouraged to use a Standardized Research Electronic Cigarette (SREC) with liquid containing 58 mg/ml nicotine for the duration of 6 weeks.
  Interventions: Other: Nicotine-Containing Electronic Cigarette
- Non-Nicotine Electronic Cigarette (Placebo Comparator): The placebo group will be provided with and encouraged to use a Standardized Research Electronic Cigarette (SREC) with liquid containing 0 mg/ml nicotine for the duration of 6 weeks.
  Interventions: Other: Non-Nicotine Electronic Cigarette

INTERVENTIONS:
Other: Nicotine-Containing Electronic Cigarette — The electronic cigarette (e-cig) used in this study will be the Standardized Research Electronic Cigarette (SREC). The SREC product is a pod-based device and comprises a replaceable pre-filled liquid reservoir ("pod") and a rechargeable power supply unit. The experimental group in this project will receive a SREC device with liquid containing 58 mg/mL of nicotine.
  Other Names: 58 mg/mL Nicotine Content SREC
  Arms: Nicotine-Containing Electronic Cigarette
Other: Non-Nicotine Electronic Cigarette — The electronic cigarette (e-cig) used in this study will be the Standardized Research Electronic Cigarette (SREC). The SREC product is a pod-based device and comprises a replaceable pre-filled liquid reservoir ("pod") and a rechargeable power supply unit. The placebo group in this project will receive a SREC device with liquid containing 0 mg/mL of nicotine.
  Other Names: 0 mg/mL Nicotine Content SREC
  Arms: Non-Nicotine Electronic Cigarette

SUMMARY:
The overall goal of this project is to understand the likely health effects of cigarette smokers switching to a Standardized Research Electronic Cigarette (SREC) and to assess the role of nicotine delivery on switching and acceptability as well as markers of health outcomes.

Current smokers who meet all eligibility criteria will completely switch from their combustible (regular) cigarettes to an electronic cigarette (SREC) that either contains 58 mg/ml of nicotine or 0 mg/ml of nicotine in the liquid.

The investigators' hypothesis is that attempting to switch to a SREC will result in a reduction in markers of harms to health, as compared with the baseline (smoking) measures. The investigators also hypothesize that nicotine-containing SRECs will facilitate switching from smoking more efficiently than zero nicotine SRECs and will result in a significantly greater improvement in markers of health risk, but will result in higher ratings of dependence on the SREC (as compared to the zero nicotine SREC).

DETAILED DESCRIPTION:
This project is a prospective parallel-group randomized double-blind, placebo-controlled study in which 104 current smokers who are willing to completely switch from their regular cigarettes to an electronic cigarette (SREC) for 6 weeks will be randomly allocated to use a SREC containing either 58 or 0 mg/ml nicotine in the liquid.

Following randomization to their assigned study product, participants will be supported in their switching efforts with regular contacts both in person at the Penn State Milton S. Hershey Medical Center and over the phone. The main measures will be recorded at two in-person visits after the randomization (switching) visit: (a) 3 weeks after switching and (b) 6 weeks after switching. All participants will also be followed up at 10 weeks by phone to identify whether they have continued to use electronic cigarettes or regular cigarettes and to assess their motivation to change.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 to 70
* Smoke ≥5 cigarettes per day for at least the past 12 months
* Smoke regular, filtered cigarettes or machine-rolled cigarettes with a filter
* Exhaled CO measurement ≥6 ppm at baseline visit
* No serious quit attempt in prior month
* Willing to completely cease cigarette consumption and switch to an e-cig
* Willing and able to attend regular visits over a 7-week period
* Able to read and write in English
* Able to understand and consent to study procedures

Exclusion Criteria:

* Unstable or significant medical condition such as COPD, kidney disease, or liver disease in the past 12 months
* Severe immune system disorders
* Women who are pregnant, trying to become pregnant, or nursing
* Use of any non-cigarette nicotine delivery product in the past 7 days
* Use of an e-cig for 5 or more days in the past 28 days or any use in the past 7 days
* Uncontrolled mental illness or substance abuse or inpatient treatment for these conditions in the past 6 months
* History of a seizure disorder or had a seizure in the past 12 months
* Currently or have ever taken medications prescribed to prevent seizures (such as Carbamazepine or Phenobarbital). Using seizure medications for off-label use (indications other than treatment for seizures) will not be included as an exclusion, these will be assessed on a case-by-case basis.
* History of difficulty providing or unwilling to provide blood samples (fainting, poor veins, anxiety, seizures)
* Surgery requiring general anesthesia in the past 6 weeks
* Use of marijuana or any illicit drug/prescription drugs for non-medical use daily/almost daily or weekly in the past 3 months per NIDA Quick Screen
* Use of hand-rolled, roll your own cigarettes
* Known allergy to propylene glycol or vegetable glycerin
* Other member of household currently participating in the study

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2022-04-22 (Actual); Primary Completion 2024-01-26 (Actual); Study Completion 2024-02-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Foulds, PhD, Principal Investigator — The Pennsylvania State University College of Medicine
Locations (1):
- The Pennsylvania State University College of Medicine, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant was excluded from the study before their assignment to a group because she did not meet the eligibility criteria for blood pressure.
Period: Randomization Period
Arm/Group | Nicotine-Containing Electronic Cigarette | Non-Nicotine Electronic Cigarette
Started | 52 | 52
Completed | 35 | 34
Not Completed | 17 | 18
Not completed — Lost to Follow-up | 7 | 12
Not completed — Withdrawal by Subject | 10 | 6
Period: 10 Week Post-treatment
Arm/Group | Nicotine-Containing Electronic Cigarette | Non-Nicotine Electronic Cigarette
Started | 35 | 34
Completed | 34 | 34
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nicotine-Containing Electronic Cigarette | Non-Nicotine Electronic Cigarette | Total
Number analyzed (Participants) | 52 | 52 | 104
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.4 (9.9) | 49.4 (9.9) | 50.9 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 33 | 68
  Male | 17 | 19 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 51 | 52 | 103
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 1 | 7
  White | 44 | 50 | 94
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 52 | 52 | 104
Education [Count of Participants; unit: Participants]
  High school or less | 11 | 9 | 20
  Greater than high school | 41 | 43 | 84

OUTCOME MEASURES:

1. Primary Outcome: Urinary NNAL Concentration
Description: Concentration of urinary carcinogen biomarker of exposure, NNAL, corrected for creatinine
Time Frame: 6-week visit (post-treatment)
Population: Four missing values because sample could not be analyzed
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Nicotine-Containing Electronic Cigarette | Non-Nicotine Electronic Cigarette
Number analyzed (Participants) | 33 | 32
ng/ml | 151.6 (235.1) | 338.2 (270.1)
Statistical Analysis 1: Comparison: Nicotine-Containing Electronic Cigarette vs Non-Nicotine Electronic Cigarette; Test type: Other; p = 0.0039, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -186.68

2. Secondary Outcome: Pulmonary Function
Description: Forced expiratory volume in one second (FEV1).
Time Frame: 6-week visit (post-treatment)
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Nicotine-Containing Electronic Cigarette | Non-Nicotine Electronic Cigarette
Number analyzed (Participants) | 35 | 34
liters | 2.7 (0.8) | 2.7 (0.8)
Statistical Analysis 1: Comparison: Nicotine-Containing Electronic Cigarette vs Non-Nicotine Electronic Cigarette; Test type: Other; p = 0.8103, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -0.06

3. Secondary Outcome: Exhaled Carbon Monoxide (CO)
Description: Exhaled CO (parts per million [ppm])
Time Frame: 6-week visit (post-treatment)
Measure: Mean (Standard Deviation); unit: ppm
Arm/Group | Nicotine-Containing Electronic Cigarette | Non-Nicotine Electronic Cigarette
Number analyzed (Participants) | 35 | 34
ppm | 10.7 (18.8) | 13.8 (11.5)
Statistical Analysis 1: Comparison: Nicotine-Containing Electronic Cigarette vs Non-Nicotine Electronic Cigarette; Test type: Other; p = 0.0105, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -3.14

4. Secondary Outcome: Urine Cotinine Concentration
Description: Cotinine (ng/ml) will serve as a measure of exposure to nicotine.
Time Frame: 6-week visit (post-treatment)
Population: Three missing values because sample could not be analyzed
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Nicotine-Containing Electronic Cigarette | Non-Nicotine Electronic Cigarette
Number analyzed (Participants) | 33 | 33
ng/ml | 5295.7 (5123.3) | 2879.7 (2481.5)
Statistical Analysis 1: Comparison: Nicotine-Containing Electronic Cigarette vs Non-Nicotine Electronic Cigarette; Test type: Other; p = 0.0182, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 2415.93

5. Secondary Outcome: Blood Pressure
Description: systolic blood pressure in mm Hg
Time Frame: 6-week visit (post-treatment)
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Nicotine-Containing Electronic Cigarette | Non-Nicotine Electronic Cigarette
Number analyzed (Participants) | 35 | 34
mmHg | 125.91 (15.74) | 124.74 (12.13)
Statistical Analysis 1: Comparison: Nicotine-Containing Electronic Cigarette vs Non-Nicotine Electronic Cigarette; Test type: Other; p = 0.8429, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 1.18

6. Secondary Outcome: Fagerstrom Test for Nicotine Dependence Mean Total Score
Description: Nicotine dependence for cigarettes will be assessed via the Fagerstrom Test for Nicotine Dependence (FTND), a measure with total scores ranging from 0 (very low dependence) to 10 (very high dependence).
Time Frame: 6-week visit (post-treatment)
Population: Questionnaire was only given to participants who used cigarettes in the past 7 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nicotine-Containing Electronic Cigarette | Non-Nicotine Electronic Cigarette
Number analyzed (Participants) | 16 | 25
score on a scale | 3.69 (2.68) | 3.2 (2.24)
Statistical Analysis 1: Comparison: Nicotine-Containing Electronic Cigarette vs Non-Nicotine Electronic Cigarette; Test type: Other; p = 0.4881, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 0.49

7. Secondary Outcome: Penn State Electronic Cigarette Dependence Index
Description: Nicotine dependence for e-cigarettes will be assessed via the Penn State Electronic Nicotine Dependence Index, a measure with total scores ranging from 0 (very low dependence) to 20 (very high dependence).
Time Frame: 6-week visit (post-treatment)
Population: Questionnaire was only given to participants who used the e-cigarette in the past 7 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nicotine-Containing Electronic Cigarette | Non-Nicotine Electronic Cigarette
Number analyzed (Participants) | 33 | 29
score on a scale | 7.21 (3.68) | 5.45 (3.47)
Statistical Analysis 1: Comparison: Nicotine-Containing Electronic Cigarette vs Non-Nicotine Electronic Cigarette; Test type: Other; p = 0.0835, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 1.76

8. Secondary Outcome: Cigarettes Per Day
Description: Mean number of cigarettes smoked per day based on the past 7 days
Time Frame: 6-week visit (post-treatment)
Population: Missing data for cigarettes per day for two participants
Measure: Mean (Standard Deviation); unit: cigarettes per day
Arm/Group | Nicotine-Containing Electronic Cigarette | Non-Nicotine Electronic Cigarette
Number analyzed (Participants) | 33 | 34
cigarettes per day | 3.78 (6.75) | 4.74 (5.21)
Statistical Analysis 1: Comparison: Nicotine-Containing Electronic Cigarette vs Non-Nicotine Electronic Cigarette; Test type: Other; p = 0.043, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -0.96

9. Secondary Outcome: Number of Participants With Abstinence From Cigarettes and Other Tobacco (Not Including E-cigs)
Description: Zero cigarettes or other tobacco products (not including e-cigs) used in the past 7 days and a CO <6ppm
Time Frame: 6-week visit (post-treatment)
Population: This is an intent-to-treat analysis so everyone who was randomized was included in the sample analyzed
Measure: Count of Participants; unit: Participants
Arm/Group | Nicotine-Containing Electronic Cigarette | Non-Nicotine Electronic Cigarette
Number analyzed (Participants) | 52 | 52
Participants | 19 | 6
Statistical Analysis 1: Comparison: Nicotine-Containing Electronic Cigarette vs Non-Nicotine Electronic Cigarette; Test type: Other; p = 0.0052, Fisher Exact; Odds Ratio (OR) = 4.35

10. Secondary Outcome: Total Score on Minnesota Nicotine Withdrawal Scale
Description: Withdrawal and craving will be assessed via the Minnesota Nicotine Withdrawal Scale. Total scores range from 0-28. Higher scores indicate worse withdrawal symptoms.
Time Frame: 1-week visit (post-treatment)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nicotine-Containing Electronic Cigarette | Non-Nicotine Electronic Cigarette
Number analyzed (Participants) | 44 | 45
score on a scale | 4.2 (4.89) | 6.16 (5.89)
Statistical Analysis 1: Comparison: Nicotine-Containing Electronic Cigarette vs Non-Nicotine Electronic Cigarette; Test type: Other; p = 0.0797, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -1.95

11. Secondary Outcome: Cigarettes Per Day
Description: Mean number of cigarettes smoked per day based on the past 7 days
Time Frame: 10-week visit (post-treatment)
Measure: Mean (Standard Deviation); unit: cigarettes per day
Arm/Group | Nicotine-Containing Electronic Cigarette | Non-Nicotine Electronic Cigarette
Number analyzed (Participants) | 34 | 34
cigarettes per day | 5.03 (8.04) | 6.47 (6.15)
Statistical Analysis 1: Comparison: Nicotine-Containing Electronic Cigarette vs Non-Nicotine Electronic Cigarette; Test type: Other; p = 0.1084, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -1.44

12. Secondary Outcome: E-cig Use Days
Description: The number of days the e-cig was used since 6-week visit (post-treatment)
Time Frame: 10-week visit (post-treatment)
Population: Data missing from participant six participants
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Nicotine-Containing Electronic Cigarette | Non-Nicotine Electronic Cigarette
Number analyzed (Participants) | 29 | 34
days | 6.69 (10.57) | 2.88 (6.84)
Statistical Analysis 1: Comparison: Nicotine-Containing Electronic Cigarette vs Non-Nicotine Electronic Cigarette; Test type: Other; p = 0.3469, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 3.81

13. Secondary Outcome: Number of Participants With Self-reported Abstinence
Description: Abstinence will be considered zero cigarettes and other tobacco products (not including e-cigs) in the past 7 days
Time Frame: 10-week visit (post-treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | Nicotine-Containing Electronic Cigarette | Non-Nicotine Electronic Cigarette
Number analyzed (Participants) | 34 | 34
Participants | 20 | 10
Statistical Analysis 1: Comparison: Nicotine-Containing Electronic Cigarette vs Non-Nicotine Electronic Cigarette; Test type: Other; p = 0.0272, Fisher Exact; Odds Ratio (OR) = 3.3632

14. Secondary Outcome: Heart Rate Variability (HRV)
Description: Heart Rate Variability (HRV) will be assessed from resting Holter EKG output.
Time Frame: 6-week visit (post-treatment)
Population: Five participants had missing data due to EKG not functioning and/or low quality data
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Nicotine-Containing Electronic Cigarette | Non-Nicotine Electronic Cigarette
Number analyzed (Participants) | 32 | 32
msec | 35.2 (17.8) | 34.6 (18)
Statistical Analysis 1: Comparison: Nicotine-Containing Electronic Cigarette vs Non-Nicotine Electronic Cigarette; Test type: Other; p = 0.589, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 0.6

15. Secondary Outcome: Presence of Premature Ventricular Contractions (PVCs)
Description: Presence of PVCs will be assessed from resting Holter EKG output.
Time Frame: 6-week visit (post-treatment)
Population: Five participants had missing data due to EKG not functioning and/or low quality data
Measure: Mean (Standard Deviation); unit: count of PVCs
Arm/Group | Nicotine-Containing Electronic Cigarette | Non-Nicotine Electronic Cigarette
Number analyzed (Participants) | 32 | 32
count of PVCs | 2 (6.8) | 2.3 (8.4)
Statistical Analysis 1: Comparison: Nicotine-Containing Electronic Cigarette vs Non-Nicotine Electronic Cigarette; Test type: Other; p = 0.5448, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -0.3

16. Secondary Outcome: ST-Elevation
Description: ST-Elevation will be assessed from resting Holter EKG output
Time Frame: 6-week visit (post-treatment)
Population: Six participants had missing data due to EKG not functioning and/or low quality data
Measure: Mean (Standard Deviation); unit: µV
Arm/Group | Nicotine-Containing Electronic Cigarette | Non-Nicotine Electronic Cigarette
Number analyzed (Participants) | 31 | 32
µV | 103.1 (97.2) | 87.8 (50.5)
Statistical Analysis 1: Comparison: Nicotine-Containing Electronic Cigarette vs Non-Nicotine Electronic Cigarette; Test type: Other; p = 0.65, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 15.3

17. Secondary Outcome: QRS Duration
Description: QRS duration will be assessed from resting Holter EKG output.
Time Frame: 6-week visit (post-treatment)
Population: Six participants had missing data due to EKG not functioning and/or low quality data
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Nicotine-Containing Electronic Cigarette | Non-Nicotine Electronic Cigarette
Number analyzed (Participants) | 31 | 32
msec | 94.3 (9.2) | 98.3 (10.4)
Statistical Analysis 1: Comparison: Nicotine-Containing Electronic Cigarette vs Non-Nicotine Electronic Cigarette; Test type: Other; p = 0.1567, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -4.0

ADVERSE EVENTS:
Time Frame: 10 weeks
Description: Adverse events (AEs) were systematically collected at each study visit by asking participants about any changes in their medication, their physical or mental health, or if they needed to seek immediate medical care at an emergency room or hospital.
Arm/Group | Nicotine-Containing Electronic Cigarette | Non-Nicotine Electronic Cigarette
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/52
Serious Adverse Events (participants affected / at risk) | 1/52 | 0/52
Other Adverse Events (participants affected / at risk) | 11/52 | 8/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nicotine-Containing Electronic Cigarette (N=52) | Non-Nicotine Electronic Cigarette (N=52)
Stroke (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nicotine-Containing Electronic Cigarette (N=52) | Non-Nicotine Electronic Cigarette (N=52)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2)
COVID-19 (Infections and infestations) | 3 (3) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-12-11): https://cdn.clinicaltrials.gov/large-docs/86/NCT03625986/Prot_SAP_000.pdf